CLINICAL TRIAL: NCT01897337
Title: The Effect of Combining Aprepitant With Ondansetron in High-risk Patients for Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yon Hee Shim, MD, PhD, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2012-0076
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant group (Experimental): We administrate aprepitant with small amount of water to aprepitant group in pre treatment room (Before patient get in the operating room)
  Interventions: Drug: Aprepitant
- placebo group (Placebo Comparator): Patient in placebo group will be given Placebo in the PTR. And we administrate ondansetron 4mg to both group 20 minutes before the end of surgery.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aprepitant — We administrate aprepitant with small amount of water to aprepitant group in pre treatment room. (Before patient get in the operating room)And we administrate ondansetron 4mg to both group 20 minutes before the end of surgery.
  Other Names: Emend
  Arms: Aprepitant group
Drug: placebo — Patient in placebo group will be given Placebo in the PTR. And we administrate ondansetron 4mg to both group 20 minutes before the end of surgery.
  Arms: placebo group

SUMMARY:
PONV (Postoperative nausea and vomiting) is one of most common complications after general anesthesia. Female sex, history of PONV, motion sickness, nonsmoker status, use of volatile agents, duration of anesthesia, opioid administration and laparoscopic surgery are known as risk factors for developing PONV. In consequence, patients undergoing laparoscopic gynecologic surgery are at high risk for developing PONV. Most of these patients use fentanyl based IV-PCA. And it also causes PONV.

So, we should prevent PONV in these patients by using multimodal or combination therapy.

Aprepitant is a NK1 receptor antagonist.And it is used to prevent chemotherapy induced nausea and vomiting. Many studies using aprepitant to prevent PONV are in progress.

In this study, we investigate the effect of combining aprepitant with ondansetron in high-risk patients for PONV.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing laparoscopic gynecologic surgery.
* Patient who takes fentanyl based IV PCA
* ASA class I-II

Exclusion Criteria:

* allergy to aprepitant
* take another antiemetics before surgery
* decreased liver function
* psychological disease
* who cannot speak Korean
* take medicines that interacts with emend who do not agree to the study

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
incidence and severity of postoperative nausea and vomiting | upto 2 days after surgery
  Severity of PONV will be measured by using verbal numerical rating scale (0-10).
  Incidence of retching or vomiting will also be recorded upto 2 days after surgery.

SECONDARY OUTCOMES:
adverse event | upto 2 days after surgery
  abdominal pain, headache, diziness, drowsiness, constipation, pruritus, etc
pain | upto 2 days after surgery
  Pain is assessed with verbal numeric rating scale. (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Yon Hee Shim, Study Director — Yonsei University
Locations (1):
- Gangnam severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Ham SY, Shim YH, Kim EH, Son MJ, Park WS, Lee JS. Aprepitant for antiemesis after laparoscopic gynaecological surgery: A randomised controlled trial. Eur J Anaesthesiol. 2016 Feb;33(2):90-5. doi: 10.1097/EJA.0000000000000242. PMID 26694939